CLINICAL TRIAL: NCT02463773
Title: Diaphragm Excursion By Ultrasound As Compared To Transpulmonary Pressure To Optimize PEEP In ARDS: A Pilot Study
Brief Title: Diaphragm Ultrasound Vs Transpulmonary Pressure To Set PEEP in ARDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Hennepin County Medical Center, Minneapolis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: G5252
Record Dates: First submitted 2015-06-02; First posted 2015-06-04 (Estimated); Results first posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-04

CONDITIONS: Acute Respiratory Distress Syndrome; Acute Respiratory Failure
Keywords: ARDS; PEEP; Critical Care Ultrasound
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ultrasound (Experimental): Adults older than 18 years old who develop ARDS, as defined by the Berlin criteria, within 72 hours of ICU admission.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Diaphragmatic excursion ultrasound assessment

SUMMARY:
This is a proof of concept study where the investigators aim to study the correlation between the use of a simple bedside ultrasound measurement of diaphragmatic muscle excursion with established (but time consuming) measurements made to optimize an important setting on the mechanical ventilator (positive end expiratory pressure or PEEP) in intubated adults with acute respiratory distress syndrome (ARDS) in the medical ICU.

DETAILED DESCRIPTION:
Ventilator induced lung injury (VILI) generates morbidity and mortality in mechanically ventilated patients. The awareness of respiratory mechanics is essential in the prevention of VILI. Currently, plateau pressures are widely used as a guide to assess alveolar pressure and minimize alveolar injury. However, patients with reduced chest wall compliance can have higher plateau pressures that may not reflect true alveolar pressure. The transpulmonary pressure has been cited as the true alveolar driving pressure because it takes into account pleural pressure that reflect chest wall mechanics; however, this requires measurement of esophageal pressure.

The investigators have experienced a disproportionate degree of excursion between the posterior and anterior right hemidiaphragm on bedside ultrasound imaging in patients with ARDS, which may reflect the dependent atelectasis that occurs during low tidal volume ventilation, cardiac weight, weight of injured lung and accumulation of extravascular lung water in critically ill patients. The optimal PEEP can be guided by measurement of esophageal pressure (and subsequent calculation of transpulmonary distending pressure) with a balloon catheter placed into the esophagus much like a nasogastric tube for enteral access. The investigators believe that the normalization of the disproportionate degree of excursion between the anterior and posterior diaphragm can also be used to identify optimal PEEP, and may be correlated with changes in transpulmonary pressure (the current gold standard).

ELIGIBILITY:
Inclusion Criteria:

* Adults older than 18 years old who develop ARDS, as defined by the Berlin criteria, within 72 hours of ICU admission.

Exclusion Criteria:

* Any contraindication for nasogastric tube placement including recent injury or pathologic condition of the esophagus.
* Major bronchopleural fistula.
* Solid organ transplant recipient.
* History or current diagnosis of diaphragmatic paralysis.
* Non-conventional mechanical ventilation strategy including high frequency oscillation, airway pressure release ventilation, prone ventilation and extra- corporeal membrane oxygenation.
* Hemodynamic instability defined as MAP<65 with multiple vasopressors.
* Declining to sign consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Prekker, MD, Principal Investigator — Hennepin County Medical Center, Minneapolis
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Cho RJ, Adams A, Ambur S, Lunos S, Shapiro R, Prekker ME. Ultrasound Assessment of Diaphragmatic Motion in Subjects With ARDS During Transpulmonary Pressure-Guided PEEP Titration. Respir Care. 2020 Mar;65(3):314-319. doi: 10.4187/respcare.06643. Epub 2019 Nov 5. PMID 31690616

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ultrasound
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ultrasound
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Feasibility
Description: This is a proof of concept study that investigates the degree of dorsal and ventral diaphragmatic excursion with bedside ultrasound during PEEP titration. Optimal PEEP management was guided by an esophageal probe calculating transthoracic pulmonary pressure. Each patient underwent a series of PEEP titrations for which data was recorded on diaphragm excursion (mm) and esophageal pressure (cmH2O). Diaphragm excursion (mm) was measured at the ventral and dorsal side using anatomic m-mode with bedside ultrasound. Esophageal pressure was measured using an esophageal probe which was placed at the bedside.
Time Frame: one year
Population: We verify that all participants met the criteria and a total of 14 were enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasound
Number analyzed (Participants) | 14
Participants | 14

ADVERSE EVENTS:
Arm/Group | Ultrasound
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes